CLINICAL TRIAL: NCT05311943
Title: Treatment With Olverembatinib in Chronic Phase Chronic Myeloid Leukemia Patients Who Failed to at Least Two Previously Administered Second-generation Tyrosine Kinase Inhibitors: a Prospective, Single-arm Clinical Trial.
Brief Title: Treatment With Olverembatinib in CML-CP Patients Who Failed to at Least Two Previously Administered Second-generation TKIs.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OLV20220331
Record Dates: First submitted 2022-03-28; First posted 2022-04-05 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-03

CONDITIONS: Olverembatinib; Chronic Myeloid Leukemia, Chronic Phase; Tyrosine Kinase Inhibitors
Keywords: olverembatinib, CML-CP
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — olverembatinib

STUDY DESIGN:
Intervention Model Description: olverembatinib, 40mg, taken orally once every other day of a 28-day cycle
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- olverembatinib (Experimental): 40mg, taken orally once every other day of a 28-day cycle
  Interventions: Drug: olverembatinib

INTERVENTIONS:
Drug: olverembatinib — olverembatinib, 40mg, taken orally once every other day of a 28-day cycle
  Other Names: HQP1351

SUMMARY:
The purpose of this trial is to evaluate the efficacy and safety of olverembatinib(HQP1351) in patients with chronic myeloid leukemia in chronic phase (CML-CP) who are resistant and/or intolerant to at least two second-generation tyrosine kinase inhibitors. The efficacy of olverembatinib is determined by evaluating the major molecular responses(MMR) at the and of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤75 years.
* Diagnosis of CML-CP.
* ECOG performance of 0-2.
* Adequate end organ function defined as the following: total bilirubin <1.5xULN, SGPT <2.5x ULN, creatinine <1.5x ULN.
* Resistance and/or intolerance of at least two second-generation TKIs.
* Patients must sign an informed consent form (ICF) indicating they are aware of the investigational nature of this study, in keeping with the policies of the hospital.

Exclusion Criteria:

* Known to be allergic to study drug ingredients or their analogues.
* History of undergone major surgery within 4 weeks.
* Patients unwilling or unable to comply with the protocol.
* Pregnant or breast-feeding patients.
* patients with other malignant tumor.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients who achieve and maintain major molecular response(MMR) at 12 months using RQ-PCR test. | 12 months
  Major molecular response (MMR) is defined as BCR-ABL1 ≤ 0.1 percent.

SECONDARY OUTCOMES:
The proportion of patients with MMR at 3, 6, 9 months. | 3, 6, 9 months.
The proportion of patients with MR 4.0 at 3, 6, 9, 12 months. | 3, 6, 9, 12 months.
  Molecular response (MR) 4.0 is defined as BCR-ABL transcripts ≤ 0.01 percent.
Proportion of patients with MR 4.5 at 3, 6, 9, 12 months. | 3, 6, 9, 12 months.
  Molecular response (MR) 4.5 is defined as BCR-ABL transcripts ≤ 0.0032 percent.
Progression free survival (PFS) | 12 months
  PFS is defined as the interval between the first dose date and the first date at which the criteria for progression are met, or death.
Overall survive (OS) | 12 months
  OS is defined as the interval between the first dose date and date of death, censored at the last contact date to be alive.
Incidence of adverse events (AEs) and serious adverse events (SAEs) to Olverembatinib. | 12 months.
  Evaluation of adverse events (AEs), serious AEs (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Xin Du, Phd, Study Chair — Shenzhen Second People's Hospital
Locations (1):
- Shenzhen Second People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No